CLINICAL TRIAL: NCT01969591
Title: Fast Track Laparoscopic Surgery: A Better Option for Treating Colorectal Cancer Than Conventional Laparoscopic Surgery
Acronym: FTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quan Wang (Other)
Responsible Party: Sponsor-Investigator, Quan Wang, Deputy Director of General Surgery, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-171; 2013-171
Record Dates: First submitted 2013-10-08; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer
Keywords: Fast track surgery, Laparoscopic surgery, colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fast-track surgery (Experimental): Patients with colorectal cancer will undergo laparoscopic colorectal resection, and will be divided into two groups. Protocols for fast-track group includes skipping preoperative mechanical bowel preparation, early restoration of diet and early postoperative ambulation.
  Interventions: Procedure: fast-track surgery
- convontional postoperative care (Other): Patients with colorectal cancer will undergo laparoscopic colorectal resection, and will be divided into two groups. Protocols for fast-track group includes skipping preoperative mechanical bowel preparation, early restoration of diet and early postoperative ambulation.
  Interventions: Other: conventional postoperative surgery

INTERVENTIONS:
Procedure: fast-track surgery — Patients with colorectal cancer will undergo laparoscopic colorectal resection, and will be divided into two groups. Protocols for fast-track group includes skipping preoperative mechanical bowel preparation, early restoration of diet and early postoperative ambulation.
  Arms: fast-track surgery
Other: conventional postoperative surgery — Patients with colorectal cancer will undergo laparoscopic colorectal resection, and will be divided into two groups. Protocols for fast-track group includes skipping preoperative mechanical bowel preparation, early restoration of diet and early postoperative ambulation.
  Arms: convontional postoperative care

SUMMARY:
To compare the outcomes of fast track laparoscopic surgery and conventional laparoscopic surgery.

DETAILED DESCRIPTION:
Method: This study is a blinded randomized trial. 70 patients with colorectal cancer will undergo laparoscopic colorectal resection, and will be divided into two groups. Protocols for fast-track group includes skipping preoperative mechanical bowel preparation, early restoration of diet and early postoperative ambulation. Outcome measures, length of hospital stay, postoperative surgical stress response (C reactive protein) and postoperative complications will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤75 years
* Good nutrition
* no systemic infection
* Elective laparoscopic surgery

Exclusion Criteria:

* Age >75 years
* Malnutrition or an organ system infection
* Associated with obstruction, bleeding, emergency surgery or surgical intervention
* Tumor with extensive metastasis
* Before operation patient was fasting, underwent gastrointestinal decompression and received nutritional support
* Previous history of abdominal surgery
* Patient had previously undergone gastrostomy

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | with the first 30 days(plus or minus 3days) after surgery
Postoperative days | with the first 30 days(plus or minus 3days) after surgery
First flatus time | with the first 30 days(plus or minus 3days) after surgery
First defecation time | with the first 30 days(plus or minus 3days) after surgery
solid diet time | with the first 30 days(plus or minus 3days) after surgery

SECONDARY OUTCOMES:
Analgesics | with the first 30 days(plus or minus 3days) after surgery
CRP (mg/L) | with the first 30 days(plus or minus 3days) after surgery
Complications:anastomotic leakage,intestinal obstruction,wound infection | one year